CLINICAL TRIAL: NCT06813261
Title: A Randomized, Placebo-Controlled, Double-Blind, Parallel-Group Pilot Trial Investigating the Impact of a Glycation Lowering (GLYLO) Supplement on Geroscience Outcomes in Postmenopausal Women
Brief Title: GLYLO Supplement Pilot Trial on Glycation and Aging in Postmenopausal Women
Acronym: GRACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Buck Institute for Research on Aging (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: BUCK_2501
Record Dates: First submitted 2025-01-13; First posted 2025-02-06 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Postmenopause; Metabolism; Geroscience
Keywords: Dietary supplement; Healthy aging; Women's health; Hormones; Advanced glycation end products (AGEs); Glycation stress; Metabolic stress

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLYLO (Experimental): a commercially available combination of glycation-lowering compounds that are GRAS (generally recognized as safe) by the FDA.
  GLYLO Ingredients Benfotiamine (fat-soluble Vitamin B1 derivative)-100mg Vitamin B6 (Pyridoxine Hydrochloride)-50mg Nicotinamide-200mg Alpha Lipoic Acid-150mg Piperine-10mg For the first week, one GLYLO capsule daily, 5 minutes after the first meal. From week 2 onwards, two capsules of GLYLO daily, one capsule after the first meal and a second capsule after the last meal.
  Interventions: Other: GLYLO
- Placebo (Placebo Comparator): Visually matched capsule with microcrystalline cellulose as an inert ingredient.
  For the first week, one placebo capsule daily, 5 minutes after the first meal. From week 2 onwards, two capsules of the placebo daily, one capsule after the first meal and a second capsule after the last meal.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: GLYLO — commercially available combination of glycation-lowering compounds that are GRAS (generally recognized as safe) by the FDA.
  GLYLO Ingredients Benfotiamine (fat-soluble Vitamin B1 derivative)-100mg Vitamin B6 (Pyridoxine Hydrochloride)-50mg Nicotinamide-200mg Alpha Lipoic Acid-150mg Piperine-10mg
  For the first week, one GLYLO capsule daily, 5 minutes after the first meal. From week 2 onwards, two capsules of GLYLO daily, one capsule after the first meal and a second capsule after the last meal.
  Arms: GLYLO
Other: Placebo — Visually matched capsule with microcrystalline cellulose as an inert ingredient.
  For the first week, one placebo capsule daily, 5 minutes after the first meal. From week 2 onwards, two capsules of the placebo daily, one capsule after the first meal and a second capsule after the last meal.
  Arms: Placebo

SUMMARY:
The aim of this study is to assess the effectiveness of GLYLO, a dietary supplement, in postmenopausal women aged 45 to 65 who are overweight or obese and have elevated HbA1c levels. Specifically, the study seeks to evaluate whether GLYLO can reduce advanced glycation end products (AGEs) levels, which are harmful compounds formed when sugar attaches to proteins or fats in the body and can contribute to aging and disease. The primary outcome of the study is to determine if GLYLO reduces AGEs, enhances metabolic and hormonal health, and mitigates age-related functional decline.

This study includes one screening visit and three testing visits over a 6-month period. After eligibility is confirmed, participants will be randomly assigned to one of two groups to take either GLYLO (two capsules daily) or a placebo at home for 24 weeks. Participants will provide blood samples at every visit. During the three testing visits, they will complete physical performance and cognitive function tests, provide both blood and urine samples, and fill out quality of life and 24-hour dietary intake questionnaires. The dietary intake questionnaires will be completed only twice i.e. at the baseline visit and again at the final 6-month visit.

DETAILED DESCRIPTION:
Telephone Screening: Subjects are screened for eligibility by telephone for major exclusion criteria. They then attend a screening visit. Eligible participants will receive an Informed Consent Form to review prior to the in-person screening visit.

Pre-Visit Requirements for all Visits: Fasting (water only) ≥10 hours, no alcohol, exercise, or cannabis products ≥10 hours.

Visit 1: Screening Visit

Upon arrival, participants will provide written consent before study procedures. A fasting blood sample will be collected for blood chemistry, hematology, lipid profile, HbA1c, and thyroid panel analysis. Participants will undergo measurements of height, weight, BMI, vital signs (blood pressure, heart rate, body temperature), and menopausal status. Medical history, current medications/supplements, and inclusion/exclusion criteria will be recorded. Eligibility will be confirmed within 2 weeks following a review by medical officers.

Visit 2: Baseline Visit Participants will undergo assessments of weight, waist/hip circumference, BMI, body composition (BIA), and vital signs. A fasting blood sample will be drawn for blood chemistry, hematology, lipids, HbA1c, and hormone panels (FSH, LH, E2, progesterone, testosterone). Additional blood will be stored for future analysis (MGO, AGEs, metabolomics, inflammation, phenotypic age). Participants will provide a midstream urine sample for archiving.

Physical Tests: Short Physical Performance Battery (SPPB), 6-minute walk test, handgrip strength.

Cognitive Tests: Montreal Cognitive Assessment (MoCA), Digit Symbol Substitution Task, Trails A & B.

Functional Tests: Skin autofluorescence (AGE Reader, DiagnOptics), Pulse Wave Velocity (PWV), retinal imaging.

Quality of life questionnaires: Pittsburgh Sleep Quality Index (PSQI), European Quality of Life 5 Dimensions (EQ-5D-5L).

Participants will receive GLYLO capsules for 12 weeks and instructions for use. They will also be provided with access to the Automated Self-administered 24-hour Dietary Assessment Tool (ASA24) and a wearable actigraphy device (Fitbit) to track activity.

At-Home Procedures Participants will take one capsule of GLYLO per day after their first meal for the first week, and two capsules per day from Week 2 onwards (after the first and last meals). They will complete a daily Study Log for 14 days, tracking product intake and symptoms. From Day 15, an abbreviated version will be used. Compliance will be monitored through telephonic interviews at Weeks 2, 4, 6, 8, 10, 14, 18, and 22. ASA24 diet logs will be completed during Weeks 1 and 23.

Visit 3: Interim Visit (3-Month Visit) Participants will return unused products and complete all assessments from the Baseline Visit. Compliance will be reviewed, and participants will receive GLYLO for an additional 12 weeks and a new Study Log.

Visit 4: Final Visit (6-Month Visit) Participants will return unused products and repeat all assessments from the Baseline and Interim Visits. They will not receive additional study products at this visit. Participants will be asked to guess the treatment they received to assess blinding.

ELIGIBILITY:
Inclusion Criteria:

1. Adults identified as female at birth with ovaries present (self-report)
2. Post menopause >1y since last menses (self-report)
3. Aged 45 - 65 y
4. Anthropometric criteria (either of the following must be met):

   * BMI ≥ 25 kg/m², based on self-reported weight and height
   * OR Waist circumference ≥88 cm, based on self-measured values. Participants may provide average home weight measurements over two consecutive days if their BMI at the screening visit is slightly below 25 kg/m².
5. HbA1c 5.5- 6.4% (screening measurement)
6. Able to read and speak English well enough to provide informed consent and understand instructions.
7. Able to attend in-person visits at The Buck Institute

Exclusion Criteria:

1. Surgical menopause (self-report)
2. Hysterectomy and/or ovariectomy (self-report)
3. Receiving systematic hormone replacement therapy (HRT) (self-report). Use of local vaginal estrogen therapy (e.g., estrogen creams, vaginal tablets, or estrogen rings such as Estring) is permitted.
4. Currently prescribed or received weight loss medications within the past 6 months or currently enrolled in a defined weight loss program. Weight must be stable (> 4%) within the last 3 months.
5. Regular use of GLYLO, or regular use of a supplement containing any of the ingredients in GLYLO, within the last 3 months.
6. Diabetes, T1DM or T2DM (self-report and screening tests): Treatment with any hypoglycemic agents (self-report), fasting glucose >125 mg/dL (screening test; may reassess once), current use of hypoglycemic drugs for non-diabetic reasons (self-report).
7. Elevated blood pressure readings (screening test): Resting Systolic Blood Pressure (SBP) ≥180 mmHg or resting Diastolic Blood Pressure (DBP) ≥100 mmHg. If a participant's blood pressure is elevated at the screening visit but not consistent with this threshold, they may provide home blood pressure readings (twice daily for two consecutive days) for the study team to evaluate eligibility.
8. Psychotropic and/or other medications known to significantly impact weight unless on a stable dose for ≥ 6 months (self-report).
9. Liver enzyme tests (alanine transaminase, aspartate transaminase) (screening test): >2 times the laboratory upper limit of normal. Reassessment during screening may be allowed under some conditions (e.g., recent use of acetaminophen).
10. Immunosuppressive disorders, taking immunosuppressive medications (including oral prednisone >10mg/day and biological immunosuppressants), or receiving chemotherapy.
11. Active gastrointestinal bleeding, or active bleeding diathesis (or resolved within 6 months prior to randomization) (self-report)
12. Active peptic ulcer disease (or resolved within 6 months prior to randomization) (self-report)
13. Active malignancy (or resolved within 6 months prior to randomization), except non-melanoma skin cancer not undergoing treatment (self-report).
14. Active infection (or resolved within 1 month prior to randomization) (self-report)
15. Allergy or hypersensitivity to any component of the supplement (self-report)
16. History of hyperthyroidism or thyroid cancer(self-report), current abnormal thyroid function (blood test at screening).
17. Cognitive status: Unable to provide informed consent to participate in and safely complete the protocol, as based on the judgment of the investigators (screening visit)
18. Psychiatric status: any condition that might affect the ability to comply with the protocol in the opinion of the Clinical Investigator or Medical Officer (screening visit)
19. Active eating disorders (self-report).
20. Active diagnosis of Gout (self-report)
21. Any change to prescription medications within 3 months prior to randomization that are judged by the study physician to impact the results of the study (self-report)
22. No overnight hospitalization within 1 month prior to randomization (self-report)
23. The presence of a condition or abnormality that in the opinion of the Investigator or Medical Officer would compromise the safety of the patient or the quality of the data

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Methylglyoxal (MGO) | Baseline, Week 12, Week 24
  MGO is a reactive dicarbonyl compound, measured by biochemical assays such as high-performance liquid chromatography (HPLC) or liquid chromatography-mass spectrometry (LC-MS) . The concentration of MGO is quantified to assess its role in the formation of advanced glycation end products (AGEs). Change is measured across the study
Advance glycation end products (AGE) | Baseline, Week 12, Week 24
  Measurement of circulating and tissue-bound AGE will be measure by either HPLC or LC-MS. Change is measured across the study

SECONDARY OUTCOMES:
Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | Baseline, Week 12, Week 24
  This is calculated by the formula HOMA-IR = (Fasting Insulin * Fasting Glucose) / 405, using fasting glucose and insulin levels. It is a marker of insulin resistance, reflecting metabolic health. Change is measured across the study
HbA1c | Baseline, Week 12, Week 24
  HbA1c is measured through immunoassay techniques, indicating average blood glucose levels over the previous 2-3 months, which is a crucial marker for long-term glucose control. Change is measured across the study
Body fat | Baseline, Week 12, Week 24
  Bioelectrical impedance analysis (BIA) is used to assess body composition, measuring fat mass. BIA calculates resistance and reactance, allowing for an estimate of body fat and lean tissue. Change is measured across the study
Body mass index (BMI) | Baseline, Week 12, Week 24
  Calculation of BMI by dividing weight (kg) by height (m²). Change is measured across the study
Hip circumference | Baseline, Week 12, Week 24
  Hip circumference is measured using a flexible tape measure, usually in centimeters, to assess fat distribution and identify central obesity, which is a risk factor for metabolic and cardiovascular diseases. Change is measured across the study
Follicle-stimulating hormone (FSH) | Baseline, Week 12, Week 24
  FSH levels are measured using immunoassays such as ELISA or radioimmunoassay, which quantify the concentration of this hormone in the blood to assess ovarian function and reproductive aging. Change is measured across the study
Muscle mass | Baseline, Week 12, Week 24
  Bioelectrical impedance analysis (BIA) is used to assess body composition, measuring lean muscle mass. BIA calculates resistance and reactance, allowing for an estimate of body fat and lean tissue. Change is measured across the study
Waist circumference | Baseline, Week 12, Week 24
  Waist circumference is measured using a flexible tape measure, usually in centimeters, to assess fat distribution and identify central obesity, which is a risk factor for metabolic and cardiovascular diseases. Change is measured across the study

OTHER OUTCOMES:
Retinal age | Baseline, Week 12, Week 24
  Retinal age is estimated using non-invasive retinal imaging techniques, such as optical coherence tomography (OCT) or fundus photography, and assessed via image analysis tools to estimate biological age based on retinal features. Change is measured across the study
Pulse wave velocity (PWV) | Baseline, Week 12, Week 24
  PWV is measured non-invasively using devices that record the speed of the blood pressure wave traveling through arteries, typically using applanation tonometry or oscillometric techniques. This reflects arterial stiffness and cardiovascular health. Change is measured across the study
Skin autofluorescence for measuring AGEs | Baseline, Week 12, Week 24
  Skin autofluorescence will be measured using the AGE Reader, DiagnOptics, which emits light at specific wavelengths and measures the amount of fluorescence emitted from the skin, correlating with AGE accumulation in tissues. Change is measured across the study
Metabolomic analysis | Baseline, Week 12, Week 24
  Comprehensive profiling of metabolites in blood is conducted using LC-MS to identify biomarkers associated with metabolic health. Change is measured across the study
Short Physical Performance Battery (SPPB) | Baseline, Week 12, Week 24
  SPPB includes tests for balance, gait speed, and chair stands. It is a composite score based on performance in these tasks consolidated to one score. Lower scores indicating poorer lower extremity function and higher frailty risk. Change is measured across the study
Hand Grip Strength | Baseline, Week 12, Week 24
  Measured in both hands using a dynamometer, which quantifies the force exerted by an individual's hand and forearm muscles. This measure is used to assess overall muscle strength and risk of frailty. Change is measured across the study
Montreal Cognitive Assessment (MOCA) | Baseline, Week 12, Week 24
  A cognitive screening tool designed to detect mild cognitive impairment and early dementia by assessing various cognitive domains. Results in a single MoCA score. Change is measured across the study
Trailmaking task | Baseline, Week 12, Week 24
  Neuropsychological test measuring visual attention, task switching, and processing speed to evaluate executive function. Change is measured across the study
Pittsburg Sleep Quality Index (PSQI) | Baseline, Week 12, Week 24
  Questionnaire about sleep quality including factors such as sleep duration, disturbances, and daytime dysfunction. A higher score reflects poorer sleep quality. Change is measured across the study
Quality of Life Questionnaire (EQ-5D-5L) | Baseline, Week 12, Week 24
  EQ-5D-5L is a standardized questionnaire assessing health-related quality of life. It includes domains like mobility, self-care, and pain, with responses used to generate a health utility score. Change is measured across the study
Ovarian hormones | Baseline, Week 12, Week 24
  Ovarian hormones are measured through blood tests using immunoassays such as ELISA or radioimmunoassays to assess hormonal levels, reflecting metabolic and reproductive aging. Change is measured across the study
Concentration of inflammatory proteins | Baseline, Week 12, Week 24
  Inflammatory biomarkers are measured in blood using immunoassays to evaluate systemic inflammation and immune response. Change is measured across the study
Phenotypic age | Baseline, Week 12, Week 24
  Calculation of biological age based on a composite of blood-based biomarkers that predict aging-related outcomes. This measure provides an estimate of physiological aging and overall health risk. Change is measured across the study

CONTACTS AND LOCATIONS:
Locations (1):
- The Buck Institute for Research on Aging, Novato, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yang DH, Chiang TI, Chang IC, Lin FH, Wei CC, Cheng YW. Increased levels of circulating advanced glycation end-products in menopausal women with osteoporosis. Int J Med Sci. 2014 Mar 13;11(5):453-60. doi: 10.7150/ijms.8172. eCollection 2014. PMID 24688308
- [Background] Merhi Z. Advanced glycation end-products: pathway of potentially significant pathophysiological and therapeutic relevance for metabolic syndrome in menopausal women. J Clin Endocrinol Metab. 2014 Apr;99(4):1146-8. doi: 10.1210/jc.2013-4465. Epub 2014 Feb 3. No abstract available. PMID 24491162
- [Background] Chaudhuri J, Bains Y, Guha S, Kahn A, Hall D, Bose N, Gugliucci A, Kapahi P. The Role of Advanced Glycation End Products in Aging and Metabolic Diseases: Bridging Association and Causality. Cell Metab. 2018 Sep 4;28(3):337-352. doi: 10.1016/j.cmet.2018.08.014. PMID 30184484